CLINICAL TRIAL: NCT05051280
Title: Combination of Cone Beam Computed Tomography and Cardiac Computed Tomography Angiography: Left Atrial Appendage Occlusion Under Three-dimensional Computed Tomography Fusion Image Guidance
Brief Title: Left Atrial Appendage Occlusion Under Cone-beam Computed Tomography Fusion Image Guidance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBCT-FIG-LAAO
Record Dates: First submitted 2021-09-12; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBCT guidance group (Experimental): Left atrial appendage occlusion under cone-beam computed tomography fusion image guidance
  Interventions: Procedure: cone-beam computed tomography fusion image

INTERVENTIONS:
Procedure: cone-beam computed tomography fusion image — Left Atrial Appendage Occlusion Under Cone-beam Computed Tomography Fusion Image Guidance

SUMMARY:
Left atrial appendage occlusion is being widely recommended as a treatment strategy for patients with nonvalvular AF to prevent stroke, especially those who cannot tolerate long-term oral anticoagulation or have other reasons for nonpharmacologic therapy. Currently, there are a number of guidance for left atrial appendage occlusion, such as transesophageal echocardiography, intracardiac echocardiogram, fluoroscopy, computed tomographic/computed tomographic angiography and so on. Procedures such as atrial septal puncture, device size selection and operational view are guided by different methods in various centers. Our center has developed a new approach to guidance: Cone-beam CT and cardiac computed tomographic angiography were combined by three-dimensional - three-dimensional image fusion in guiding left atrial appendage occlusion.

DETAILED DESCRIPTION:
Eligible NVAF patients were recruited consecutively and received our LAAO workflow of local anesthesia, intracardiac echocardiography-guided transseptal puncture, and 3DCTA-3DCBCTF fusion-guided occluder implantation. The primary outcome was optimal occluder implantation (successful implantation with no occluder recapture and replacement). Other outcomes were procedure/fluoroscopic time, contrast agent consumption, radiation dose, and peri-procedure complications. We compared our results with existing publications of LAAO guided by 3DCTA and two-dimensional fluoroscopy (3DCTA-2DF) fusion images.

ELIGIBILITY:
Inclusion Criteria:

1. An age of >18 years;
2. A CHA2DS2-VASc score of ≥2;
3. Clinical conditions allowing TEE and sedation;
4. Left ventricular ejection fraction >30%;
5. And at least one of the following indications: (a) HAS-BLED score of ≥3; (b) intolerance to long-term OAC, and (c) stroke, transient ischemic attack, or thromboembolism even under oral anticoagulation treatment;

Exclusion Criteria:

1. A glomerular filtration rate of <50 mL/min/1.73 m2;
2. The presence of a thrombus in the LA and LAA;
3. Acute myocardial infarction or unstable angina, decompensated heart failure (New York Heart Association functional class III-IV), or heart transplantation;
4. Stroke or transient ischemic attack within 30 days;
5. Very poor peripheral vessel access not allowing device delivery;
6. Moderate or massive pericardial effusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of success at first device selected | In surgery
  successful occluder deployment and release with no being resized

CONTACTS AND LOCATIONS:
Overall Officials: JUN PU, Doctor, Study Chair — Shanghai Jiao Tong University, School of Medicine, Affiliated Ren Ji Hospital
Locations (1):
- Shanghai Jiaotong University School of Medcine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No